CLINICAL TRIAL: NCT05116891
Title: A Phase 1 / 2 Study of CAN04, a Fully Humanized Monoclonal Antibody Against IL1RAP, in Combination With Different Chemotherapy Regimens in Subjects With Advanced Solid Tumours
Brief Title: A Phase 1/2 Study of CAN04 in Combination With Different Chemotherapy Regimens in Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cantargia AB (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAN04CLIN004
Record Dates: First submitted 2021-10-07; First posted 2021-11-11 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Advanced Solid Tumors; Colorectal Cancer; Non Small Cell Lung Cancer; Biliary Tract Cancer
Keywords: Nadunolimab; CAN04; CRC; NSCLC
MeSH Terms: conditions — Colorectal Neoplasms; Carcinoma, Non-Small-Cell Lung; Biliary Tract Neoplasms | interventions — Oxaliplatin; Fluorouracil; Leucovorin; Docetaxel; Gemcitabine; Cisplatin

STUDY DESIGN:
Intervention Model Description: Dose Escalation Phase (Phase 1):
  mFOLFOX and Gemcitabine/Cisplatin Arm: Subjects with any type of locally advanced or metastatic cancer who have no therapeutic alternatives with proven survival benefit or who are eligible for mFOLFOX or gemcitabine/cisplatin (G/C) backbone chemotherapy as standard of care (SoC) for the next-line treatment.
  Docetaxel Arm: Subjects with locally advanced or metastatic non-small cell lung cancer (NSCLC) cancer who have no therapeutic alternative with proven survival benefit or who are eligible for docetaxel (DTX) backbone chemotherapy as SoC for the next-line treatment.
  Phase 2: Subjects with locally advanced or metastatic colorectal cancer (mCRC), NSCLC, or biliary tract cancer (BTC) who are eligible for mFOLFOX, DTX, or G/C treatment, respectively.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CAN04 and chemotherapy (mFOLFOX) (Experimental): 12 cycles for mFOLFOX/CAN04-Each cycle is 2 weeks.mFOLFOX/CAN04 treatment arm: CAN04 and mFOLFOX are administered on Day 1 with a mFOLFOX continuation of regime on Day 2. CAN04 is only administered on Day 1.
  Interventions: Drug: CAN04 (nadunolimab); Drug: mFOLFOX
- CAN04 and chemotherapy (DTX) (Experimental): 6 cycles for DTX/CAN04, Cycles are 3 weeks. DTX/CAN04 treatment arm: CAN04 and DTX are administered on Day 1 followed by CAN04 in monotherapy on Day 8.
  Interventions: Drug: CAN04 (nadunolimab); Drug: DTX
- CAN04 and chemotherapy (G/C) (Experimental): 8 cycles for G/C/CAN04, Cycles are 3 weeks. G/C/CAN04 treatment arm: CAN04 and G/C are administered on Day 1/Day 8.
  Interventions: Drug: CAN04 (nadunolimab); Drug: G/C

INTERVENTIONS:
Drug: CAN04 (nadunolimab) — FULLY HUMANISED MONOCLONAL ANTIBODY AGAINST IL1RAP
  Other Names: nadumolimab
Drug: mFOLFOX — mFOLFOX/CAN04
  Other Names: Modified Folfox; Oxaliplatin, 5-fluorouracil (5-FU), leucovorin
  Arms: CAN04 and chemotherapy (mFOLFOX)
Drug: DTX — DTX/CAN04
  Other Names: Docetaxel
  Arms: CAN04 and chemotherapy (DTX)
Drug: G/C — G/C/CAN04
  Other Names: Gemcitabine and cisplatin
  Arms: CAN04 and chemotherapy (G/C)

SUMMARY:
This is a Phase 1/2, open-label, multicentric, non-randomised, parallel-arm study that aims to establish the safety, tolerability, and initial efficacy of CAN04 in combination with 3 SoC chemotherapies (mFOLFOX, DTX, and G/C).

ELIGIBILITY:
Inclusion Criteria:

PHASE 1 and PHASE 2:

* Subject must be able to understand and sign written informed consent, according to local guidelines.
* Subject must be ≥18 years of age at the time of signature of the ICF.
* Subject must have an ECOG PS score of 0 or 1.
* Subject must have adequate organ function, as indicated by the laboratory values in the protocol
* Women of childbearing potential must have a negative serum pregnancy test before study entry. Women of non-childbearing potential will have had at least 24 continuous months of natural (spontaneous) amenorrhea, and an appropriate clinical profile (eg, age appropriate, history of vasomotor symptoms), or have had hysterectomy, bilateral salpingectomy or bilateral oophorectomy>6 weeks before screening.
* Male or female subjects: Male subjects with female partners of childbearing potential and female subjects of childbearing potential are required to use 2 forms of acceptable contraception, including 1 barrier method, during their participation in the study and for 4 months after the last dose of CAN04 or for 6 months after the last dose of the relevant chemotherapies, whatever is longer. Male subjects must also refrain from donating sperm during their participation in the study and in the period when contraceptives are required
* Subjects must not have contraindications according to the approved local summary of product characteristics (SmPC) for the respective components of the SoC chemotherapies.

PHASE 1 (Dose Escalation)

* Subject has histologically or cytologically confirmed diagnosis of locally advanced cancer or metastatic cancer. Subjects do not need to have measurable disease per response evaluation criteria in solid tumours (RECIST) v1.1.
* Subject has a condition where all standard therapeutic options with proven survival benefit have been exhausted, refused by the subject, or are contraindicated. OR Subject has a condition where 1 of the 3 study regimens (mFOLFOX, DTX, or G/C) is considered SoC for the next-line treatment.
* Subject has additional disease characteristics per treatment arm:

  * mFOLFOX Arm: All subjects eligible for mFOLFOX can be enrolled. A maximum of 2 previous lines of cytotoxic chemotherapy treatment for metastatic disease is allowed (targeted agents without cytotoxic effect will not be counted).
  * DTX Arm: Subjects eligible to receive DTX as monotherapy for NSCLC can be enrolled in this treatment arm. No more than 2 lines of prior systemic anti-cancer therapies for the metastatic disease are allowed. Targeted therapy is not counted as prior therapy. Subjects who received DTX monotherapy in a prior line of therapy are not eligible.
  * G/C Arm: All subjects eligible for G/C can be enrolled (including first-line treatments).. Subjects with BTC will be prioritized.

PHASE 2 All treatment arms in Phase 2 (CRC, NSCLC or BTC)

* Subject must have at least 1 measurable lesion as defined by RECIST v1.1. Tumour lesions that have been irradiated ≥4 weeks before the start of treatment, and have subsequently had documented progression, may be chosen as target lesions in the absence of measurable lesions that have not been irradiated.
* Only applicable after the second interim analysis has been performed: Primary or metastatic lesion amenable to biopsy and willingness of the subject to undergo a screening (if no adequate archival tissue is available) and an on-treatment biopsy (as defined in the protocol). The lesion accessible for biopsy may not be the only target lesion and should not be located in a previously irradiated field (unless this index lesion has PD ≥20% after radiation). The requirement(s) for the screening and/or on-treatment biopsy and/or archival tissue may be waived by the sponsor for individual sites and subjects, in particular if tumour locations are not safely accessible, after discussion and documented agreement between the site and the sponsor´s medical monitor.

CRC Arm

* Subject has definitive histologically or cytologically confirmed metastatic or locally advanced adenocarcinoma of the colon or rectum without possibility of locoregional treatment with curative intention or candidate for curative metastasectomy
* Subject has received at least 2 prior lines of therapy for non-resectable locally advanced or metastatic CRC and has progressed or is intolerant to those therapies. If the tumour is microsatellite instability-high, it should have progressed on a previous immune CPI unless contraindicated, or such therapy is not available to the subject. Subjects with KRAS wildtype should be eligible to receive mFOLFOX and should have received anti-EGFR therapy unless contraindicated or not available for the subject.
* Note: For subjects who received adjuvant or neoadjuvant chemotherapy and had recurrence within 6 months of completion of the adjuvant or neoadjuvant chemotherapy, the adjuvant or neoadjuvant therapy is counted as the first line of chemotherapy for the metastatic disease.

NSCLC Arm

* Subject has histologically or cytologically confirmed squamous or non-squamous NSCLC unresectable stage IIIB/C or stage IV for whom monotherapy DTX treatment is indicated.
* Subject received platinum-based therapy and a programmed cell death protein 1 or programmed death-ligand 1 inhibitor as prior treatment regimens (unless contraindicated or such therapy is not available to the subject). Prior CPIs and chemotherapy may have been administered alone or in combination. No more than 2 prior lines of cytotoxic chemotherapy containing regimens for the advanced or metastatic disease are allowed.

Note: Subjects who received DTX monotherapy in a prior line of therapy are not eligible.

* Subjects who received adjuvant or neoadjuvant chemotherapy and had recurrence within 6 months of completion of the adjuvant or neoadjuvant chemotherapy are allowed to count the adjuvant or neoadjuvant therapy as the first line of chemotherapy for the recurrent/metastatic disease.
* Subject eligible for mutation-targeted therapies (eg, osimertinib, alectinib, crizotinib, larotrectinib, capmatinib, pralsetinib) must have exhausted treatment options for targeted therapies available locally

BTC Arm

* Subject has histopathological or cytological biliary tract carcinoma (intrahepatic or extrahepatic cholangiocarcinoma, gallbladder cancer, or ampullary carcinoma) non-resectable, recurrent, or metastatic amenable for G/C treatment indicated as SoC.
* Subject has not received standard systemic anti-cancer therapies neither for non-resectable locally advanced nor for metastatic disease.
* Note: Subjects who received adjuvant or neoadjuvant chemotherapy and had recurrence within 6 months after completion of the adjuvant or neoadjuvant chemotherapy are eligible for the study.

Exclusion Criteria:

* Subject has a known or suspected allergy to study drugs (including chemotherapy regimens), any of its components.
* Subject has another histologically confirmed cancer different from those described in inclusion criteria, except for cervical carcinoma in situ, superficial non-invasive bladder tumour, curatively treated stage I non-melanoma skin cancer, or prostate cancer subjects curatively treated with surgery or radiation and not receiving systemic or androgen deprivation therapy. Subjects with a history of another cancer, different from that described in the inclusion criteria, can be enrolled if the cancer was curatively treated ≥5 years ago and non-recurrence has been documented in the past 2 years.
* Subject has uncontrolled or significant heart failure defined as New York Heart Association Classification III or IV.
* Subjects to receive mFOLFOX or DTX: having peripheral sensory neuropathy Grade ≥2.
* Subject has QT interval corrected using Fridericia's formula (QTcF) >480 msec at screening.
* Subjects to receive DTX and CAN04: if they have liver metastases and aspartate aminotransferase (AST) and/or ALT >1.5 × upper limit of normal (ULN) concomitant with alkaline phosphatase >2.5 × ULN.
* Subject has uncontrolled brain metastases. Subjects are allowed to be enrolled if brain metastasis has been previously treated with surgery, and/or stereotactic radiosurgery and are considered controlled (controlled by the dose ≤10 mg/day of prednisone or equivalent) at the time of the first dose of CAN04. For asymptomatic subjects, without known brain metastases, brain imaging during screening is not required. Subjects with known brain metastases should have undergone brain imaging in the frame of the imaging screening procedures.
* Subject has an active severe infection requiring parenteral antibiotics at the time of enrolment or subjects currently receiving oral antibiotics as a continuation of a previous course of parenteral antibiotics. Subjects can be enrolled when antibiotic treatment is complete and if there are no signs of residual infection. Note: Subjects with BTC who required stent placement should have the procedure completed 2 weeks before and be free of antibiotics (oral or parenteral) for at least 1 week before first treatment administration.
* Subject has a history of a relevant autoimmune disease as per assessment of the investigator or autoimmune disease requiring systemic immunosuppressive therapy (daily prednisone equivalent doses >10 mg/day).
* Subject is expected to require any other form of systemic or localised anti-neoplastic therapy while on study (including maintenance therapy with another agent, radiation therapy, and/or surgical resection).
* Subject has had an allogeneic tissue/solid organ transplant.
* Subject received a live vaccination, etanercept, or other tumour necrosis factor-alpha inhibitors prior to (within 28 days of first study drug administration) participation in this study. For severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) vaccines, a wash-out of 2 weeks before first administration of study drug is recommended.
* Subject had treatment with systemic anti-cancer treatments, or major surgery within 4 weeks before the first dose of study drug or 5 half-lives, whichever is shorter. Subjects should have recovered from previous treatment toxicity to Grade 1, baseline (except alopecia and peripheral neuropathy).
* Subject received radiotherapy ≤4 weeks before the start of treatment (≤2 weeks for palliative irradiation to peripheral tumour lesions, other than for example spine or pelvis, without increased risk for delayed cytopenias) and has not recovered to Grade 1 or better from related toxicity of such therapy (except for alopecia).
* Subject has known hepatitis B virus surface antigen seropositive or detectable hepatitis C infection viral load. Note: Subjects who have positive hepatitis B core antibody or hepatitis B surface antigen antibody can be included but must have an undetectable hepatitis B viral load.
* Subjects who test positive for human immunodeficiency virus (HIV) are NOT excluded from this study but must meet the following criteria:

  * Have cluster of differentiation 4 (CD4)+ T-cell (CD4+) counts ≥350 cells/μL.
  * Have not had an opportunistic infection within the past 12 months. Subjects on prophylactic anti-microbials can be included in the study.
  * Should be on established anti-retroviral therapy for at least 4 weeks.
  * Have an HIV viral load less than 400 copies/mL before enrolment.
* Subject has a known history of any other relevant congenital or acquired immunodeficiency other than HIV infection.
* Subject has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Subject has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study.
* Subject has any medical condition, co-morbidity, physical examination finding, metabolic dysfunction, or clinical laboratory abnormality that, in the opinion of the investigator, renders the subject unsuitable for participation in a clinical study due to high safety risks and/or potential to affect interpretation of results of the study.
* Subject has known allergy to any of the drugs or excipients in the allocated treatment.
* Only subjects in the G/C arm: Subjects who, as per applicable local label, due to hearing impairment or ongoing phenytoin administration, have contraindication for cisplatin.

mFOLFOX Arm/CRC Arm Exclusion Criteria

* Subjects with clinical laboratory test values at screening below the lower limit of normal for any of the following electrolytes: potassium, magnesium, corrected or ionised calcium.

  * NOTE: Subjects achieving normal values for these electrolytes with supplements during the screening period are allowed at the discretion of the investigator. Serum chemistry documenting normal electrolyte values is required prior to each dose of oxaliplatin.
* Subjects with congenital long QT syndrome or a history of ventricular arrhythmias, including bradyarrhythmia (<50 beats per minute).
* Subjects with existing uncompensated heart disease: myocardial ischaemia or early (up to 4 weeks) post-infarction status, congestive heart failure, left ventricular hypertrophy, cardiomyopathy, conduction disorder within 6 months before enrolment.
* Subjects with dihydropyrimidine dehydrogenase (DPD) deficiency or who have been treated within 4 weeks of first dose of study treatment with potent DPD inhibitors (eg, brivudine, sorivudine). Subjects who previously received 5-FU without toxicity that can be correlated with DPD deficiency do not need to be tested
* Subjects with pernicious anaemia or other anaemias due to vitamin B12 deficiency that cannot be corrected before the first dose of mFOLFOX.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-09-22 (Actual); Primary Completion 2023-06-23 (Actual); Study Completion 2023-06-23 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of CAN04 in combination with selected standard hemotherapy regimens and to establish MTD and/or RP2D. | Until 30 days after the last dose of study treatment (EOT visit) in Phase 1
  Frequency, duration, and severity of AEs
To assess the preliminary efficacy of CAN04 in combination with chemotherapy regimens measured as tumour response. | Until approximately 3 years after last treatment in Phase 2.
  ORR defined as the percentage of subjects with PR or CR based on RECIST v1.1.

SECONDARY OUTCOMES:
To assess preliminary anti-tumour activity of CAN04 in combination with selected standard chemotherapy regimens. | Every 12 weeks until disease progression or death from any cause in Phase 1.
  ORR/iORR, PFS/iPFS according to RECIST v1.1/iRECIST 1.1 DCR/iDCR measured as a percentage of subjects with CR/iCR + PR/iPR + SD/iSD ≥16 weeks Duration of response (DOR)
To assess preliminary anti-tumour activity of CAN04 in combination with selected standard chemotherapy regimens. | Until approximately 3 years after last treatment in Phase 2.
  iORR, PFS/iPFS according to RECIST v1.1/iRECIST 1.1 DCR/iDCR measured as a percentage of subjects with CR/iCR + PR/iPR + SD/iSD ≥16 weeks Duration of response (DOR) Overall Survival (OS)
To further characterise the safety and tolerability of CAN04 in combination with chemotherapy at the MTD/RP2D. | Until 30 days after the last dose of study treatment (EOT visit) in Phase 2.
  Frequency, duration, and severity of AEs
To assess preliminary anti-tumour activity of CAN04 in combination with selected standard chemotherapy regimens. | Until 30 days after the last dose of study treatment (EOT visit).
  Change from baseline upon treatment in serum biomarkers: CEA and CA19-9 (CEA for subjects with CRC; CEA and CA19-9 for subjects with BTC), Changes from baseline upon treatment in ECOG, PS and body weight
To assess PK of CAN04 after a single dose and at steady state | From first dose until 30 days after the last dose of study treatment (EOT visit)
  Serum concentrations of CAN04

OTHER OUTCOMES:
To evaluate the effect of CAN04 when administered in combination with chemotherapy on subject-reported cancer-related fatigue. | Until 30 days after the last dose of study treatment (EOT visit) in Phase 2
  Changes upon treatment in Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Scores.
To evaluate the effect of CAN04 when administered in combination with chemotherapy on health-related quality of life. | Until 30 days after the last dose of study treatment (EOT visit) in Phase 2
  Changes upon treatment in European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30 scores
To assess changes in serum biomarker IL-6 when CAN04 is administered in combination with standard of care chemotherapy. | From first dose until 30 days after the last dose of study treatment (EOT visit).
  Changes in serum concentration of IL-6.
To assess changes in serum biomarker IL-8 when CAN04 is administered in combination with standard of care chemotherapy. | From first dose until 30 days after the last dose of study treatment (EOT visit).
  Changes in serum concentration of IL-8.
To assess changes in serum biomarker CRP when CAN04 is administered in combination with standard of care chemotherapy. | From first dose until 30 days after the last dose of study treatment (EOT visit).
  Changes in serum concentration of C-reactive protein (CRP).
To assesschanges in serum biomarker sILRAP when CAN04 is administered in combination with standard of care chemotherapy. | From first dose until 30 days after the last dose of study treatment (EOT visit).
  Changes in serum concentration of soluble IL1RAP.
To assess ADA formation against CAN04. | Until 30 days after the last dose of study treatment (EOT visit).
  ADA against CAN04

CONTACTS AND LOCATIONS:
Overall Officials: Ignacio Garcia-Ribas, MD, PhD, Study Director — Cantargia AB
Locations (6):
- France (4):
  - EDOG Institut de Cancerologie de l'Ouest - PPDS, Saint-Herblain, Boulevard Jacques Monod
  - Centre Georges François Leclerc, Dijon, Côte-d'Or
  - Institut Bergonie, Bordeaux
  - Centre Eugene Marquis, Rennes
- Spain (2):
  - Hospital Universitari Vall D'Hebron, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid

IPD SHARING:
Plan to Share IPD: No